CLINICAL TRIAL: NCT01189032
Title: Dose-Response Study of DE-089 Ophthalmic Solution in Patients With Dry Eye -Late Phase II Confirmatory Study-
Brief Title: Late Phase II Confirmatory Study of DE-089 Ophthalmic Solution in Patients With Dry Eye
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Santen Pharmaceutical Co., Ltd. (Industry)
Other Study IDs: 00890404
Record Dates: First submitted 2010-08-24; First posted 2010-08-26 (Estimated); Results first posted 2014-08-08 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

ARMS (3):
- High concentration (Experimental)
  Interventions: Drug: DE-089 ophthalmic solution
- Low concentration (Experimental)
  Interventions: Drug: DE-089 ophthalmic solution
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo ophthalmic solution

INTERVENTIONS:
Drug: DE-089 ophthalmic solution
  Arms: High concentration
Drug: DE-089 ophthalmic solution
  Arms: Low concentration
Drug: Placebo ophthalmic solution
  Arms: Placebo

SUMMARY:
Dose response related to efficacy and safety of DE-089 ophthalmic solution are examined in patients with dry eye, using a multicenter, randomized, double-blind, parallel group comparison study, and the optimal concentration is determined.

ELIGIBILITY:
Inclusion Criteria:

* Those who show:

  * Keratoconjunctival disorder confirmed with vital dye staining
  * Abnormal Schirmer score results

Exclusion Criteria:

* Eye disease that needs therapy other than that for dry eye
* Those who need to wear contact lenses during the clinical study

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Primary Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Santen study sites, Osaka, Osaka, Japan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Excluded (n=34)
Groups:
- Placebo: Placebo ophthalmic solution
- Low Concentration: 1% DE-089 ophthalmic solution
- High Concentration: 3% DE-089 ophthalmic solution
Period: Overall Study
Arm/Group | Placebo | Low Concentration | High Concentration
Started | 94 | 96 | 96
Completed | 89 | 89 | 90
Not Completed | 5 | 7 | 6
Not completed — Adverse Event | 1 | 3 | 4
Not completed — Lack of Efficacy | 2 | 3 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Protocol Violation | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Low Concentration | High Concentration | Total
Number analyzed (Participants) | 94 | 96 | 96 | 286
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (17.3) | 57.9 (16.3) | 56.4 (17.8) | 56.6 (17.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 85 | 77 | 238
  Male | 18 | 11 | 19 | 48

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Fluorescein Staining Score From Baseline
Description: Fluorescein staining was scored according to the protocol by Shimmura et al. The cornea was divided into 3 equal zones: upper, middle, and lower. Each zone had a staining score ranging between 0 and 3 points, with minimum and maximum total staining scores ranging between 0 and 9 points. 0 is better.
  The degree of staining with Fluorescein dyes was scored as follows: 0 = no staining, 1= staining of less than half of the area, 2= staining of more than half of the area, 3= staining in the whole area.
Time Frame: Baseline and 4-week (discontinued(LOCF))
Population: Efficacy analysis was performed per protocol set (PPS). Excluded cases were 7 subjects (3 subjects in 3% group, 3 subjects in 1% group, and 1 subject in Placebo group).
  The reason of exclusion: used the prohibited concomitant drug, dosing period shortage, number of doses non-compliance, or had no available efficacy data.
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Placebo | Low Concentration | High Concentration
Number analyzed (Participants) | 93 | 93 | 93
points | -0.95 (1.33) | -1.34 (1.43) | -1.55 (1.30)
Statistical Analysis 1: Comparison: Placebo vs Low Concentration vs High Concentration; Test type: Superiority or Other; p = 0.004, maximum contrast method — It's the p-value of linear trend. It's adjusted for multiplicity; To confirm dose-response relation, two contrasts were provided; linear trend (-1, 0, 1), and saturated at 1% DE-089 ophthalmic solution (-2, 1, 1)
Statistical Analysis 2: Comparison: Placebo vs Low Concentration vs High Concentration; Test type: Superiority or Other; p = 0.006, maximum contrast method — It's the p-value of Saturated at 1% DE-089. It's adjusted for multiplicity; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Arm/Group | Placebo | Low Concentration | High Concentration
Serious Adverse Events (participants affected / at risk) | 0/94 | 0/96 | 1/96
Other Adverse Events (participants affected / at risk) | 17/94 | 14/96 | 28/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=94) | Low Concentration (N=96) | High Concentration (N=96)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 — There was a serious adverse event in 3% DE-089 ophthalmic solution group.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=94) | Low Concentration (N=96) | High Concentration (N=96)
Eye irritation (Eye disorders) | 3 | 7 | 13
Eye pain (Eye disorders) | 4 | 2 | 6
Nasopharyngitis (Infections and infestations) | 10 | 5 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No